CLINICAL TRIAL: NCT02692937
Title: Is Chronic Whiplash-associated Pain of Neurogenic Origin? A Study Protocol of a Randomized Controlled Trial Comparing Neurolysis of Peripheral Nerves With Traditional Neck-specific Exercise
Brief Title: Is Chronic Whiplash-associated Pain of Neurogenic Origin?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Project no 6168/2207
Record Dates: First submitted 2016-02-15; First posted 2016-02-26 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Whiplash Injuries
Keywords: Neurosurgical Procedures; Nerve Block; Exercise therapy; Physical Therapy Specialty
MeSH Terms: conditions — Whiplash Injuries | interventions — Nerve Block

ARMS (2):
- Surgery and exercise (Experimental): Neurolysis of peripheral nerves in the back of the head and/or neck. Traditional neck-specific exercise program including five individual treatments sessions within 3 months plus home program over 9 months.
  Interventions: Procedure: Neurolysis; Other: Traditional neck-specific exercise program
- Exercise, Active Comparator (Active Comparator): Traditional neck-specific exercise program including five individual treatments sessions within 3 months plus home program over 9 months.
  Interventions: Other: Traditional neck-specific exercise program

INTERVENTIONS:
Procedure: Neurolysis
  Arms: Surgery and exercise
Other: Traditional neck-specific exercise program

SUMMARY:
The purpose of this study is to compare the effects of neurolysis with the effects of a exercise program on pain and other symptoms in individuals with chronic whiplash (WAD II-III).

DETAILED DESCRIPTION:
People with whiplash associated disorders (WAD) grade II-III have chronic severe pain and symptoms and reduced quality of life. The origin of the symptoms is still unknown, and there are to date no available guidelines for treatment of this condition. The lack of effective treatment leads to high costs for the patients, and to society, due to considerable medical care and work loss.

After providing a written consent, the patients will be randomized to either surgical treatment with neurolysis of peripheral nerve/s in the back of the head and/or neck plus physiotherapy or to physiotherapy (care-as-usual) only. Both groups will be treated with the same traditional neck-specific exercise program for 12 months. All participants will be evaluated with patient-reported outcomes and clinical examination at baseline, and at 6, 12 and 24 months after inclusion.

The main outcome will be change in NDI from baseline to the 2-year follow-up. A preliminary sample-size calculation shows that 27 patients are needed for each treatment arm to detect a clinically important change of 10 points in NDI, with a between-group standard deviation of 13 point (statistical power of 80 % and a 5% significance level). To account for a 20% drop-out rate, 32 patients will be included per arm. Because this is the first RCT on neurolysis vs care-as-usual treatment, a second sample-size calculation including empirical data will performed by an independent statistician, without breaking the code, when 30 patients in each group have been included. Secondary outcomes include VAS (average pain including pain in the head, neck and face), symptom index, self-efficacy, HDI, WAD-DI, psychosomatic aspects, quality of life and clinical examination. Data will be performed with parametric, or non-parametric statistics, as appropriate, in IBM SPSS Statistics version 22 for Mac (IBM Corp., Armonk, NY, USA). Analysis will be performed according to both intention-to-treat and per protocol. To account for missing data, the previous group means value will be considered to remain form the last occasion and used as carry forward. For continuous data, differences in mean change (baseline vs follow-up) will be compared between groups and adjusted in relation to baseline values. For categorical data, differences in median change (baseline vs follow-up) will be compared between groups and adjusted in relation to baseline values. Effect sizes will be calculated for all measures.

This Randomized Controlled Study is approved and funded by the National Board of Health and Welfare in Sweden (project no 6168/2007).

ELIGIBILITY:
Inclusion Criteria:

* trauma that has caused a whiplash injury
* at least one year of incapacitating chronic neck pain/headache related to the injury (WAD II-III)
* typical trigger points in the back of the head or in the neck and significant pain relief with local anesthesia towards the painful areas

Exclusion Criteria:

* mental illness
* abuse of drugs/alcohol
* not understanding or reading the Swedish language
* previous surgery in the back of the head

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2017-03 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The Neck Disability Index (NDI) | 24 months
  Questionnaire

SECONDARY OUTCOMES:
The Symptom index | 24 months
  Related symptoms (pain) psychosomatic aspects and any disability due to the neck complaint. Questionnaire.
Self-Efficacy Scale (SES) | 24 months
  Questionnaire
Headache Disability Index (HDI) | 24 months
  Questionnaire
Whiplash Associated Disorders - Disability Index (WAD-DI) | 24 months
  Questionnaire
Zung Self-Rating Depression Scale (Zung) | 24 months
  Questionnaire
Modified Somatic Perception Questionnaire (MSPQ) | 24 months
  Questionnaire
EuroQol questionnaire (EQ-5D) | 24 months
  Questionnaire
EuroQol thermometer (EQ-VAS) | 24 months
  Questionnaire
Cervical range of motion (CROM) | 12 months
Pain drawing, perceived face and body sensations | 12 months
  The characteristics of the patients sensations/pain are described on two different charts.
Exploratory outcome. Perceived pain on a Numeric Rating Scale (NRS) for 14 specific trigger points in the muscles of the occipital region, neck and shoulder. | 12 months
  The physiotherapist palpates each trigger point, according to a detailed protocol developed for the present study.

CONTACTS AND LOCATIONS:
Overall Officials: Leif Anderberg, MD, PhD, Principal Investigator — The Department of Neurosurgery, Skåne University Hospital
Locations (1):
- The Department of Neurosurgery, Skåne University Hospital, Lund, Skåne County, Sweden